CLINICAL TRIAL: NCT05118425
Title: A Real-world Study of the Dietary Perceptions and Practices in Chinese Psoriasis Patients
Brief Title: Dietary Perceptions and Practices in Chinese Psoriasis Patients
Status: Completed | Type: Observational
Sponsor: Xijing Hospital (Other)
Responsible Party: Principal Investigator, Gang Wang, MD, chief of dermatology, Xijing Hospital
Other Study IDs: XijingH-PF-20210220
Record Dates: First submitted 2021-10-10; First posted 2021-11-12 (Actual); Last update posted 2021-11-12 (Actual); Status verified 2021-11

CONDITIONS: Psoriasis
Keywords: Diet; psoriasis; perception; practice
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The influences of diet on psoriasis have been long discussed. As reported in previous publications, a majority of U.S. psoriasis population show high interest in the role of diet on their skin conditions. Given the distinct traditional perceptions and lifestyles in China, the dietary beliefs and behaviors in Chinese psoriasis patients would be very likely to show different patterns. Nevertheless, the information of this large population is still unknown. In this regard, the investigators conduct a questionnaire-based survey, aiming to assess the dietary perceptions and behaviors of Chinese psoriasis patients.

DETAILED DESCRIPTION:
A total of 25 medical institutions all over China participated in the survey. Psoriasis patients surveyed were from both outpatient and inpatient dermatology departments. Researchers from each institution were trained for assisting patients to fill the questionnaire. Each participant filled the online-based questionnaire anonymously in a private setting. The questionnaire consisted of 54 main questions and extended questions, concerning the profile of disease conditions, perceptions and behaviors of diet in their daily life.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old.
* Confirmed diagnosis of psoriasis.
* Duration of psoriasis ≥ 3 years.
* Must be able to read and understand the questionnaire.
* Receive a full explanation of the purpose and content of the trial before the study begins, and voluntarily sign a written consent form.

Exclusion Criteria:

* Unable to read or understand the questionnaire.
* Other conditions deemed by the investigator to be inappropriate for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The survey is a nation-wide study conducted in 25 hospitals or institutions in China, aiming to observe the dietary perceptions and practices in Chinese adult psoriasis patients. The patient population covered 31 provinces and 241 cities over China.
Sampling Method: Non-Probability Sample
Enrollment: 3453 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Practices of food choice in Chinese psoriasis patients. | Information collection: over a span of 2 months
  The cross-sectional study design consisting of a questionnaire survey. We conducted a cross-sectional study through Chinese Umer Doctor and WeChat platforms. The survey is a national program of studies aimed to evaluate the perception of nutrition in Chinese psoriasis patients over the age of 18 and its impact on disease. A total of 25 medical institutions participated in the survey, and the patient population covered 31 provinces and 241 cities. A specific self-administered questionnaire was designed for this study to be administered electronically to all patients. The questionnaire includes 54 main questions and extended questions, 15 items refer to the demographic and disease characteristics, 28 items refer to the dietary practices (eg. avoiding or adding certain food or dietary supplements), the the outcomes of the intervention, as well as factors related to different dietary practices.

SECONDARY OUTCOMES:
Perceptions of the correlation between diet choice and disease severity in Chinese psoriasis patients. | Information collection: over a span of 2 months
  10 questions in the questionnaire was designed to detect the perceptions of the influence of dietary modification in patients conducting different dietary practices and the factors related to different perceptions.

CONTACTS AND LOCATIONS:
Overall Officials: Gang Wang, Principal Investigator — Dermatology Derpartment of Xijing Hospital
Locations (1):
- Dermatology Derpartment of Xijing Hospital, Xi'an, Shaanxi, China